CLINICAL TRIAL: NCT05159505
Title: Strategies for the Implementation of an Interdisciplinary Juvenile Scoliosis Correction Program Based on ERAS Principles. Before-after Study.
Brief Title: Interdisciplinary Scoliosis Correction Program.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Jowita Biernawska, MD PhD, Pomeranian Medical University Szczecin
Other Study IDs: KB-0012/126/10/2021/Z
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Juvenile; Scoliosis; ERAS; Complication,Postoperative; Complication of Surgical Procedure
MeSH Terms: conditions — Scoliosis; Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- "the before" group: 40 teenagers after scoliosis surgery before interdisciplinary program implementation
- "the after" group 1: 40 teenagers after scoliosis surgery after ERAS program implementation
- "the after" group 2: 40 teenagers after scoliosis surgery after ERAS and educational program implementation

SUMMARY:
The aim of this study is to compare the outcomes after scoliosis surgery before and after the implementation of an interdisciplinary juvenile scoliosis correction program in teenager based on ERAS (enhanced recovery after surgery) principles.

DETAILED DESCRIPTION:
Creating an optimal protocol for interdisciplinary care in the perioperative period in terms of therapeutic management (anesthesia and surgery schedule), as well as care, rehabilitation and ensuring mental well-being determines the real impact on the reduction of the risk of complications in the perioperative period. Enhanced recovery after surgery (ERAS) protocol has been found to result in reduced lenght of stay and complications in adult patients. Data in pediatric population remains modest. In addition to ERAS principles our terapeutic team has created a special educational application for better patient preparation for surgery. The purpose of the application is to explain the general rules of conduct in the process of preparing and carrying out surgery, anesthesia, prehabilitation and physiotherapy in children undergoing orthopedics surgery (e.g. spine surgery for adolescent idiopathic scoliosis).

Hypothesis: Implementing an interdisciplinary juvenile scoliosis correction program based on ERAS principles and special educational app. will improve patient outcomes leading to a statistically significant reduction in post-operative pain and opioids demand, complication rate, length of stay without increasing readmissions and cost.

ELIGIBILITY:
Inclusion Criteria:

* patient with age < 18 years
* patient scheduled for idiopatic scoliosis surgery

Exclusion Criteria:

* patient with age > 18years others type of scoliosis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Caucasian children undergoing orthopedics surgery (e.g. spine surgery for adolescent idiopathic scoliosis).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
type of complications | up to 4 weeks after surgery
  surgery and anaesthesia complications

SECONDARY OUTCOMES:
Postoperative length of hospital stay | up to 4 weeks after surgery
  Postoperative length of hospital stay
Number of Analgetics consumption | up to 6 days after surgery
  consumption including opioids and non-opioids drug
Time to first bowel motion | up to 6 days after surgery
  Able to eat without abdominal discomfort, nausea, or vomiting
Time to first verticalization | up to 6 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided
nd